CLINICAL TRIAL: NCT03026647
Title: Evaluation of Suture Material for Closure of Hysterotomy
Brief Title: Suture Material for Closure of Hysterotomy
Status: Withdrawn | Type: Observational
Why Stopped: Not moving forward staff shortage
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, Principal Investigator, St. Louis University
Other Study IDs: 27509
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cesarean Section; Complications, Wound, Hematoma
MeSH Terms: conditions — Wounds and Injuries; Hematoma | interventions — Sutures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Suture — To examine different types of suture material used for hysterotomy closure in cesarean section and determine if one is preferred above other types due to a complications profile.

SUMMARY:
Retrospective chart review evaluating different suture types on surgical outcomes for cesarean delivery and vaginal birth after cesarean delivery outcomes when different sutures are used.

DETAILED DESCRIPTION:
Cesarean sections are one of the most common surgeries performed in the United States; approximately 1 out of 3 births are completed by cesarean delivery. In 2014, 1,284,551 cesarean deliveries were performed. Unfortunately, even with this being a very common procedure some surgical topics have not been fully evaluated. One of these topics is the choice of suture for repair of the hysterotomy (uterine) incision. Several suture materials are available, yet only polygatactin-910 and catgut have been evaluated in a single study. In this study, only surgery complications were evaluated. Catgut was found to be associated with less risk of receiving a blood transfusion, otherwise no differences were found. One of the most common suture materials used at our institution is poliglecaprone 25, however no long term studies have been completed for this indication. In addition, no studies have evaluated the risk of uterine rupture with trial of labor after cesarean after using poliglecaprone 25 to repair the hysterotomy. This information could be very useful in counseling for patients. As the cesarean delivery rates continue to climb, information on appropriate technique for surgery are needed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who underwent a cesarean delivery or vaginal birth after cesarean

Exclusion Criteria:

* unable to give consent

Ages: 14 Years to 55 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Female, pregnant, All ethnic backgrounds,
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Preferred suture | 3 months
  Preferred suture chart review

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No